CLINICAL TRIAL: NCT01780142
Title: Longitudinal Observational Study of Severe Asthma
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130059; 13-H-0059
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01-21

CONDITIONS: Asthma
Keywords: Airflow Obstruction; Corticosteroid Resistance; Exacerbations; Quality of Life; Airway Inflammation; Natural History
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- asthmatics: Subjects with confirmed diagnosis of asthma without other lung disease followed for collection of clinical data & specimens
- non-asthmatic healthy volunteers: Healthy volunteers in whom asthma has been ruled out and without other lung disease followed for comparison to asthmatics

SUMMARY:
Background:

- Asthma is a lung condition that causes difficulty breathing and decreased lung function. Some people with asthma have more severe disease symptoms. They may be less responsive to standard treatments such as steroids. Researchers want to compare severe asthmatics with mild or moderate asthmatics or people without asthma over a long period. This information may help identify new treatments for people whose asthma is not well controlled by standard medications.

Objectives:

- To compare severe asthmatics with mild or moderate asthmatics, and healthy volunteers, to study the progression and outcomes of the disease.

Eligibility:

* Individuals at least 18 years of age who have been diagnosed with asthma for at least 1 year.
* Healthy volunteers at least 18 years of age.

Design:

* This study will involve an initial visit to the NIH Clinical Center for all participants. Selected participants may be asked to return for repeat visits over a number of years. The test results from participants with asthma will be compared with those from the healthy volunteers.
* All participants will be screened with a physical exam and medical history.
* Participants may (but will not necessarily) have the following tests at each visit:
* Complete medical history and physical exam
* Blood, urine, sputum, and nasal cell samples
* Breath tests and heart and lung function tests
* Six-minute walk test to measure ability to exercise
* Imaging studies such as chest x-rays, bone density scans, and sinus scans
* Allergy skin testing
* Vocal cord exam
* Overnight sleep study
* Participants may remain on the study for as long as they are willing to participate and do not develop health problems that will interfere with the study.

DETAILED DESCRIPTION:
Asthma is a common disease and a significant public health problem, affecting one in every 10 individuals, nearly 30 million people in the US alone. About 5-10% of asthmatics have severe disease that is difficult to control with standard therapies. Severe asthmatics are considered to be relatively resistant to corticosteroids, a mainstay of therapy in asthma. Furthermore, chronic corticosteroid therapy often results in side effects that adversely affect outcomes. Thus, more effective treatment options, which are safe, cost-effective and easy to administer, are needed for severe asthmatics.

As our understanding of asthma evolves, it is becoming clearer that there are distinct phenotypes that differ regarding demographic factors such as age, sex and race, but also, perhaps more importantly, with regards to clinical, physiologic and biologic characteristics. This heterogeneity may reflect distinct pathogenic mechanisms that result in airflow obstruction and the clinical presentation of asthma. In turn, a better understanding of the different factors that contribute to disease severity and pathogenesis will be necessary to identify new, personalized treatment and management approaches for severe asthmatics. Our goal is to gain a better understanding of the pathogenic mechanisms that differentiate severe asthma from mild to moderate asthma, including the role of the above-mentioned factors on disease control. In so doing, we hope to discover novel pathways that can be manipulated to achieve our primary aim of developing new therapies for severe asthmatics.

ELIGIBILITY:
* All volunteer subjects must be at least 18 years of age and must be able to provide informed, written consent for participation in this study. Subjects will be recruited irrespective of age, sex, race or ethnicity. Eligibility in the study is determined on the basis of the following inclusion and exclusion criteria.

INCLUSION CRITERIA - ASTHMATICS:

* Subjects must be over 18 years of age.
* Subjects must have had a diagnosis of asthma, as defined by the American Thoracic Society, for at least one year to enter this study.
* Subjects must have a history of reversible airflow obstruction, as defined by a positive response to inhaled bronchodilators or a positive methacholine bronchoprovocation challenge by ATS criteria. Severe, refractory asthma will be defined by the 2000 ATS workshop consensus criteria. Refractory asthmatics will meet one or both of the major criteria and at least two minor criteria as outlined in the Protocol. This definition is applicable only to patients in whom (1) other conditions have been excluded, (2) exacerbating factors have been optimally treated, and (3) poor adherence does not appear to be a confounding issue. Compliance or medication adherence will be assessed at the initial and subsequent visits by questioning the subjects about their medication use (self-report).
* If asthmatic subjects do not fulfill the criteria for severe asthma, they will be classified as mild to moderate asthmatics.
* Subjects must have the ability to provide informed consent.

INCLUSION CRITERIA - NON-ASTHMATICS:

* Subjects must be at least 18 years of age without a clinical diagnosis of asthma.
* Subjects must have no evidence of obstructive airway disease, as defined by ATS criteria on spirometry, and a negative methacholine bronchoprovocation challenge.
* Subjects must have the ability to provide informed consent.
* Subjects will be matched to asthmatics by gender and age (+/- 10 years).

EXCLUSION CRITERIA:

* Any concurrent condition (medical, social or behavioral) that, in the opinion of the research team, would preclude or confound acquisition or interpretation of data or delivery of care.
* Subjects must not be pregnant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of subjects will be aimed at selecting our study population of interest, severe asthmatics of both genders and all races over the age of 18 years. Mild and moderately severe asthmatics, as well as age (+/- 10 years) and gender matched healthy volunteers (non-asthmatics), will be enrolled for comparison to severe asthmatics. Asthmatics with other concomitant conditions, e.g. other lung diseases such as COPD, which may confound the data collected, may be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
To collect longitudinal data regarding the natural history, co-morbid conditions, complications and outcomes of severe asthmatics as compared to mild or moderate asthmatics and non-asthmatics | all
  we hope to discover novel pathways that can be manipulated to achieve our primary aim of developing new therapies for severe asthmatics.

CONTACTS AND LOCATIONS:
Overall Officials: Amisha V Barochia, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Barochia AV, Gordon EM, Kaler M, Cuento RA, Theard P, Figueroa DM, Yao X, Weir NA, Sampson ML, Stylianou M, Choy DF, Holweg CTJ, Remaley AT, Levine SJ. High density lipoproteins and type 2 inflammatory biomarkers are negatively correlated in atopic asthmatics. J Lipid Res. 2017 Aug;58(8):1713-1721. doi: 10.1194/jlr.P077776. Epub 2017 Jun 27. PMID 28655726
- [Background] Barochia AV, Kaler M, Cuento RA, Gordon EM, Weir NA, Sampson M, Fontana JR, MacDonald S, Moss J, Manganiello V, Remaley AT, Levine SJ. Serum apolipoprotein A-I and large high-density lipoprotein particles are positively correlated with FEV1 in atopic asthma. Am J Respir Crit Care Med. 2015 May 1;191(9):990-1000. doi: 10.1164/rccm.201411-1990OC. PMID 25692941
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-H-0059.html